CLINICAL TRIAL: NCT05581836
Title: The Effect of Central Sensitization and Neuropathic Pain on Patients Reported Outcomes Following Total Knee Arthroplasty
Brief Title: The Effect of Central Sensitization and Neuropathic Pain After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Other Study IDs: KC22RASI0362
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has been well known that central sensitization (CS) is a risk factor for inferior outcomes following total knee arthroplasty (TKA). However, there are still insufficient studies on the relationship between CS and neuropathic pain (NP), and the effects of CS and NP on the patient-reported outcome measures (PROMs) of patients who underwent TKA. The purpose of this study was to investigate the relationship between CS and NP and whether CS and NP were associated with PROM in patients undergoing TKA.

DETAILED DESCRIPTION:
A total of 312 patients who underwent primary TKA for end stage knee OA were enrolled. CS was defined as a patient with a score of 40 or higher using central sensitization inventory (CSI). NP was defined as a patient with a score of 12 or more using pain detect questionnaire (PDQ). PROMs were also evaluated based on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score preoperatively and at postoperative 1 year. The patients were divided into 4 groups, group 1 with CS and NP positive, group 2 with only CS positive, group 3 with only NP positive, and group 4 with CS and NP negative, and PROM was compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee degenerative osteoarthritis
* Patients for total knee arthroplasty over the age of 60
* Patients with 2 year postoperative medical records

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Neuropsychiatric patients
* Hepatic insufficiency
* Renal insufficiency
* Allergy or intolerance to study medications
* Patients with an acetylsalicylic acid of IV (angina, congestive heart failure, dementia, cerebrovascular accident)
* Chronic opioid use (taking opioids for longer than 3 months)
* Alcohol, drug abuser
* Narcotics addiction

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study was approved by the Institutional Review Board of our hospital. Between May 2019 and February 2020, a total of 332 primary TKAs were performed at our institution by a single surgeon. Only patients with a follow-up period of more than two years were included in the study. The remaining 316 patients with primary TKAs were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | 2 years after TKA
  Western Ontario and McMaster University Arthritis Index (WOMAC) scale is a validated questionnarie for evaluation of patients who underwent knee operation. The questionnaire consists of 24 tiems, with five pain-related categories (score range 0-20), two stiffness categories (score range 0-8), and 17 physical functional categories (score range 0-68). All items were scored on a 5-point Likert scale (0 = none, 1 = slightly, 2 = moderate, 3 = serious, 4 = extreme). Total score range is 0-96. The lower the score, the better the result.

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic Univerisity of Korea Seoul St Mary's hospital, Seoul, South Korea